CLINICAL TRIAL: NCT07062055
Title: Bevacizumab Plus QL1706 Combined With Stereotactic Body Radiotherapy in Patients With BCLC Stage C Hepatocellular Carcinoma With Portal Vein Tumor Thrombus or Extrahepatic Oligometastatic Metastases (BRAVE): A Prospective, Multicenter, Single-Arm Phase II Study
Brief Title: BRAVE Study: QL1706 + Bevacizumab + SBRT for BCLC-C HCC With PVTT or Oligometastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinbo Yue, Director of Radiation Oncology Department, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2025-152-02
Record Dates: First submitted 2025-06-24; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma; Portal Vein Tumor Thrombus; Oligometastases; Radiotherapy; Immunotherapy; Anti-VEGF Therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Immunotherapy; Hyperthermia, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Drug: Bevacizumab (15 mg/kg, IV, every 3 weeks) Drug: QL1706 (7.5 mg/kg, IV, every 3 weeks, administered sequentially after bevacizumab) Radiation: Stereotactic Body Radiotherapy (SBRT), total dose of 25-50 Gy in 5 fractions over 1-2 weeks, targeting intrahepatic tumors, portal vein tumor, and/or limited extrahepatic oligometastatic lesions
  Interventions: Drug: Anti-VEGF; Drug: Immunotherapy; Radiation: Local Therapy

INTERVENTIONS:
Drug: Anti-VEGF — Drug: Bevacizumab (15 mg/kg, IV, every 3 weeks)
Drug: Immunotherapy — QL1706 (7.5 mg/kg, IV, every 3 weeks, administered sequentially after bevacizumab)
Radiation: Local Therapy — Stereotactic Body Radiotherapy (SBRT), total dose of 25-50 Gy in 5 fractions over 1-2 weeks, targeting intrahepatic tumors, portal vein tumor, and/or limited extrahepatic oligometastatic lesions

SUMMARY:
This multicenter, prospective, single-arm Phase II clinical trial is designed to evaluate the efficacy and safety of combining bevacizumab and QL1706 with stereotactic body radiotherapy (SBRT) in patients with Barcelona Clinic Liver Cancer (BCLC) stage C hepatocellular carcinoma (HCC) who present with portal vein tumor thrombus (PVTT) or extrahepatic oligometastatic disease. The study aims to determine whether this combination strategy can prolong progression-free survival (PFS), while also improving overall survival (OS), objective response rate (ORR), disease control rate (DCR), and duration of response (DoR), as well as maintaining quality of life (QoL). In addition, the trial will systematically evaluate the safety profile and treatment-related toxicities associated with this regimen.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) remains a major clinical challenge, primarily due to its frequent diagnosis at advanced stages and the limited proportion of patients eligible for curative surgical interventions. For individuals with advanced or unresectable disease, current treatment options include targeted therapy, immunotherapy, and radiotherapy. Although these modalities have led to incremental improvements in survival outcomes, the overall prognosis remains unsatisfactory, with only modest gains in progression-free survival (PFS) and overall survival (OS).

Among systemic therapies, multi-targeted tyrosine kinase inhibitors (TKIs) such as sorafenib and lenvatinib have been widely adopted as first-line treatments. However, their clinical benefits are limited by low objective response rates (ORR), significant adverse events, and the eventual emergence of drug resistance. In light of these limitations, anti-angiogenic agents such as bevacizumab have emerged as promising alternatives. Bevacizumab not only inhibits tumor angiogenesis but also modulates the tumor microenvironment to enhance antitumor immune responses, offering a potential synergistic effect when combined with immune checkpoint inhibitors (ICIs).

QL1706 is a novel bispecific antibody targeting both programmed cell death protein 1 (PD-1) and cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), designed to enhance T cell-mediated antitumor immunity through dual immune checkpoint blockade. Compared to conventional monoclonal antibodies, this dual-targeting strategy may offer improved antitumor efficacy without a proportional increase in immune-related toxicity. Preliminary clinical studies across multiple tumor types have demonstrated a favorable safety and efficacy profile, supporting its potential for broader oncologic application. Moreover, emerging preclinical and early-phase clinical data suggest that the combination of QL1706 and bevacizumab may have particular therapeutic synergy in HCC.

Stereotactic body radiotherapy (SBRT) is a highly precise radiation technique capable of delivering ablative doses to tumor lesions while sparing surrounding healthy tissue. In patients with HCC who are ineligible for surgical resection, SBRT has shown promising outcomes in terms of local tumor control and overall survival. Beyond its cytotoxic properties, SBRT may enhance tumor immunogenicity by promoting antigen release and modulating the tumor microenvironment, thereby potentiating the effects of immunotherapy.

This prospective, multicenter, single-arm Phase II clinical trial is designed to evaluate the efficacy and safety of a combination regimen comprising bevacizumab, QL1706, and SBRT in patients with Barcelona Clinic Liver Cancer (BCLC) stage C HCC with portal vein tumor thrombus (PVTT) or extrahepatic oligometastatic disease. The primary endpoint is PFS. Secondary endpoints include OS, ORR, disease control rate (DCR), duration of response (DoR), quality of life (QoL), and safety, as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

Exploratory analyses will investigate immunologic responses and biomarker dynamics, including programmed death-ligand 1 (PD-L1) expression, immune cell infiltration (e.g., CD8⁺T cells, natural killer cells), and vascular endothelial growth factor (VEGF)-related alterations within the tumor microenvironment. Patient-reported outcomes, including health-related quality of life, will be assessed using validated instruments such as the EORTC QLQ-C30 questionnaire.

ligible patients are required to provide written informed consent and must meet all inclusion criteria as confirmed by imaging and pathological evaluation. The treatment regimen consists of bevacizumab, QL1706, and SBRT. SBRT will be delivered to the intrahepatic primary tumor, PVTT, and any identified extrahepatic oligometastatic lesions.

This combination strategy maximizes antitumor efficacy by integrating three complementary mechanisms of action: anti-angiogenesis, immune activation, and localized tumor ablation. Through comprehensive clinical, radiologic, and biomarker-based assessments, this trial aims to determine whether such a multimodal therapeutic approach can provide meaningful clinical benefit for patients with BCLC stage C HCC complicated by PVTT or extrahepatic oligometastatic disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged between 18 and 70 years.
2. Histologically confirmed or clinically diagnosed HCC based on the 2024 Guidelines for Diagnosis and Treatment of Primary Liver Cancer issued by the National Health Commission of the People"s Republic of China.
3. BCLC stage C disease, with either PVTT and/or extrahepatic oligometastases. Oligometastases are defined as≤5 metastatic lesions involving≤3 organs.
4. Liver function classified as Child-Pugh class A or B (score≤7).
5. At least one measurable lesion according to RECIST v1.1: defined as a lesion with a longest diameter >1.5 cm, or ≥1 lesion with a longest diameter >1.0 cm and at least two perpendicular diameters measurable.
6. ECOG performance status score ≤2.
7. Expected survival time ≥3 months.
8. Adequate organ function (liver, kidney, lung, and heart) to tolerate both local radiotherapy and systemic therapy.
9. Patients of reproductive potential must agree to use reliable contraception during the study and for at least 12 months after the end of treatment.
10. Ability to understand and voluntarily sign written informed consent prior to initiation of any study-specific procedures.

Exclusion Criteria:

1. Presence of a second primary malignancy.
2. BCLC stage C patients not meeting the criteria for oligometastases.
3. Presence of brain metastases or peritoneal carcinomatosis.
4. PVTT or metastatic lesions not amenable to radiotherapy.
5. Prior chemotherapy or systemic anticancer therapy.
6. Severe impairment of liver, kidney, lung, or cardiac function that would preclude tolerating radiotherapy or systemic treatment.
7. Serious medical comorbidities that may interfere with study participation, including but not limited to uncontrolled diabetes, active peptic ulcer disease, or other significant cardiopulmonary conditions (as judged by the investigator).
8. Severe or uncontrolled infections, or active autoimmune diseases.
9. Neurological disorders affecting central nervous system function.
10. Pregnant or breastfeeding women, or women of childbearing potential not using effective contraception.
11. Known allergy or hypersensitivity to any of the study drugs.
12. Patients deemed unsuitable for the study for any other reason at the discretion of the investigator.thrombus (PVTT), and/or limited extrahepatic lesions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2028-07-25 (Estimated); Study Completion 2029-07-25 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Two years
  The time between enrollment and disease progression or death for patients in the intent-to-treat population, whichever occurred first; for those who did not progress at the time of withdrawal from the study or whose time to disease progression was not recorded, the date of the last visit was used as the endpoint date.

SECONDARY OUTCOMES:
Overall Survival (OS) | Five years
  Time from initiation of treatment to death from any cause.
objective response rate (ORR) | Two years
  The proportion of patients whose tumor size decreases (partial response) or disappears (complete response) after radiation based on RECIST 1.1.
Disease Control Rate (DCR) | Two years
  The proportion of patients whose tumor size decreases (partial response), disappears (complete response), or is stable after radiation based on RECIST 1.1.
Duration of Response (DoR) | Two years
  The time in patients whose tumor size decreases (partial response), disappears (complete response), or is stable after radiation based on RECIST 1.1.
Incidence of Treatment-related adverse events | Five years
  Treatment-related adverse events will be assessed and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Specific examples of expected toxicities include, but are not limited to:
  Gastrointestinal disorders: Abdominal distension (visible or palpable enlargement of the abdomen); Abdominal pain; Belching; Subjective sensation of gastric bloating or fullness; Nausea (with or without retching or urge to vomit); Vomiting; Dyspepsia (characterized by burning sensation, bloating, nausea, or discomfort); Constipation; Diarrhea; Dysphagia (difficulty in swallowing); Upper gastrointestinal bleeding General disorders and administration site conditions: Fatigue; Pain, such as radiation-associated pain at sites of bone metastases or liver region pain Respiratory disorders: Dyspnea (shortness of breath); Radiation pneumonitis Skin and subcutaneous tissue disorders: Radiation dermatitis.
Change in Quality of Life Assessed by EORTC QLQ-C30 Questionnaire | Two years
  Quality of life will be assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). Changes from baseline to follow-up time points will be analyzed across multiple domains including physical, emotional, and social functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Jinbo Yue, Doctor, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No